CLINICAL TRIAL: NCT00279253
Title: Effects of Intravenous Clonidine on Ocular Blood Flow and Intraocular Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-141003
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2006-01

CONDITIONS: Physiology
Keywords: clonidine; glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Clonidine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: clonidine (drug) intravenously

SUMMARY:
Background Clonidine, a derivate of Imidazol, is an antihypertensive drug. It acts by stimulating adrenergic receptors on nerves in the brain and Imidazol-receptors. As a result, clonidine slows the heart rate and reduces blood pressure. Clonidine was approved by the FDA in 1974 and is registered in Austria with the brand name "Catapresan".

Alpha2 adrenergic agonists are nowadays used topically as eye drops in glaucoma treatment. In addition to their known effect of lowering intraocular pressure, alpha2 adrenoceptor agonists are neuroprotective. Brimonidine, which is the most commonly used topical alpha-2 agonist, is currently on the market for treatment of glaucoma and is effective in reducing intraocular pressure. It has, however, been shown that brimonidine is a very potent vasoconstrictor in the ciliary body thus reducing aqueous humor production. Little is, however, known about potential vasoconstrictor effects of brimonidine in the posterior pole of the eye. This is of clinical importance, because optic nerve head ischemia appears to contribute to glaucoma pathophysiology. Direct investigation of the ocular hemodynamic effects of brimonidine is, however, difficult, because lowering intraocular pressure with brimonidine may confound the results due to the concomitant change in ocular perfusion pressure.

The aim of the present study is to assess the effect of intravenous clonidine as model drug of alpha agonists on ocular blood flow and IOP in healthy humans.

Study objectives:

To investigate effects of clonidine on ocular blood flow and intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

Men aged between 19 and 35 years, nonsmokers

Body mass index between 15th and 85th percentile

Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant

Normal ophthalmic findings, ametropy < 3 Dpt.

Exclusion Criteria:

Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study

Treatment in the previous 3 weeks with any drug

Symptoms of a clinically relevant illness in the 3 weeks before the first study day

History of hypersensitivity to the trial drug or to drugs with a similar chemical structure

History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs

Blood donation during the previous 3 weeks

History or family history of epilepsy

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2004-03; Study Completion 2005-01

PRIMARY OUTCOMES:
ocular blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, MD, Principal Investigator — Department of Clinical Pharmacology